CLINICAL TRIAL: NCT00282490
Title: Sacral Transcutaneous Nerve Stimulation Treatment for Functional Daytime Incontinence in Children With Over Active Bladder Syndrome
Brief Title: Surface Nerve Stimulation Treatment for OAB in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHTENS2006; 2006-41-6085,; 20050180
Record Dates: First submitted 2006-01-25; First posted 2006-01-26 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: Overactive bladder; Children; Nerve stimulation; TENS
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Nerve stimulator

SUMMARY:
The purpose of this study is to perform a randomized controlled investigation of the effect of surface nerve stimulation on functional daytime incontinence in children with OAB.

DETAILED DESCRIPTION:
Daytime urinary incontinence is common in children. At the age of 7 a prevalence of 2-9 % has been reported. Daytime urinary incontinence is a heterogenic multifactorial illness where the the symptoms has several degrees of severity and can be caused by different mechanisms. Daytime urinary incontinence can be etiologically classified in the rare neurogenic and structural forms and the common functional or idiopathic form (where no neurological or structural cause of the bladder dysfunction can be identified.

The symptom based diagnosis OAB (overactive bladder) is most often used to describe daytime urinary incontinence in children. OAB is defined as a symptom syndrome including urgency with or without urge incontinence in combination with frequency.

When urinary tract infection and neurogenic and structural causes has been excluded the nonpharmacological bladder rehabilitation is first line treatment of OAB. It is expected that approximately 50 % of the children can be relieved of symptoms by this treatment. In the non-responding cases behavioural modifying regimes can be coupled with anticholinergic medication. However, poor compliance of the child or parents, or dose limiting side effects often influences the efficacy of this intervention. Also a considerable number of children experience no or only limited effect from the treatment even though all instructions are complied with. This has let to research into new treatment modalities and the use of low frequency electrical current to inhibit detrusor overactivity in adults has become common. Pilot studies have indicated a significant effect of TENS on urinary incontinence in children with OAB.

Hypothesis:

* Sacral TENS is an effective treatment of urinary incontinence in children with OAB refractory to anticholinergic medication coupled with bladder training and voiding reeducation.
* The acute effect of sacral TENS can be identified by urodynamics
* It is possible to predict the outcome of sacral TENS treatment in these children.

  30 children (age 5-14 years) with functional daytime incontinence refractory to anticholinergic medication coupled with bladder training. The study protocol consists of 1 week of basic home registrations and a 4 day in-patient phase succeeded by a 4 week home training period. The participants will be randomized to treatment with either active or inactive TENS.

ELIGIBILITY:
Inclusion Criteria:

* Daytime urinary incontinence with at least 1 episode of at least 1 ml per week
* Incontinence refractory to treatment
* Informed consent

Exclusion Criteria:

* Severe diseases of the kidneys or urinary tract besides OAB

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Clinical effects evaluated by home registrations of degree of incontinence, VAS score of degree of urgency and frequency volume charts at specified intervals. Acute effect evaluated by urodynamics.

SECONDARY OUTCOMES:
Bladder capacity, voiding frequency and subjective impression of incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Hagstroem, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of pediatrics,Skejby Sygehus, University hospital of Aarhus, Aarhus, Aarhus N, Denmark